CLINICAL TRIAL: NCT04470570
Title: The Effects of Cross-Education and Blood Flow Restriction Study on Patients Undergoing Shoulder Arthroscopy
Brief Title: The Effect of Cross-Education on Shoulder Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Michael Banffy, MD, Director, Orthopedic Sports Medicine Fellowship, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000737
Record Dates: First submitted 2020-07-07; First posted 2020-07-14 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Injuries; Rotator Cuff Repair
Keywords: biceps tenodesis; Cross-Education; Blood-Flow Restriction Training
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): This group will undergo a standardized rehabilitation protocol of the involved shoulder only.
- Cross-Education Group (Experimental): This group will undergo a standardized rehabilitation protocol of the involved shoulder with the addition of upper extremity strengthening exercises to the uninvolved side.
  Interventions: Other: Cross-Education
- Cross-Education + Blood-Flow Restriction Group (Experimental): This group will undergo a standardized rehabilitation protocol of the involved shoulder with the addition of upper extremity strengthening exercises to the uninvolved side with blood-flow restriction simultaneously.
  Interventions: Other: Cross-Education; Other: Blood-Flow Restriction Training

INTERVENTIONS:
Other: Cross-Education — 1) Cross-Education: The effect that exercising the uninvolved upper extremity will have a positive effect on the involved upper extremity.
  Arms: Cross-Education + Blood-Flow Restriction Group; Cross-Education Group
Other: Blood-Flow Restriction Training — 1) Blood Flow Restriction: A type of resistance training using a blood-pressure like cuff that partially occludes venous blood flow to induce various neurohormonal effects and allows strength gains to be achieved at very low loads of resistance.
  Arms: Cross-Education + Blood-Flow Restriction Group

SUMMARY:
The purpose of this study is to examine the effectiveness of a strength training protocol on the uninjured upper extremity either alone or with the addition of blood flow restriction (BFR) training on subjects who have undergone shoulder arthroscopy.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effectiveness of a strength training protocol on the uninjured limb either alone or with the addition of blood flow restriction (BFR) training on the status of the injured limb post shoulder arthroscopy. Patients will be randomized into one of three standardized physical therapy (PT) groups after shoulder arthroscopy: Control group (CON), Strength Training on the uninvolved shoulder (STR), strength training with the BFR on the uninvolved shoulder (BFR). All three patient groups will follow a standardized PT rehab protocol that is usual standard of care on the involved shoulder. The STR and BFR group will follow a typical standard of care rehab protocol to the uninvolved side to investigate the potential effects of cross-education. Isometric strength will be assessed utilizing handheld dynamometry (HHD) at Kerlan-Jobe during their regularly scheduled pre-operative and follow-up visits. Patients age 18 and older undergoing shoulder arthroscopy for rotator cuff repair and/or biceps tenodesis. The study includes 3 visits which are standard of care pre-operative and post-operative visits. The duration of the study will be 14 weeks. 2 weeks to allow for a pre-op baseline strength assessment and 12 weeks post-op for the final assessment during the patients routine follow-up visit. Physical Therapy will be standardized for all three groups in terms of frequency and rehabilitation protocol. The only exercises that will be added will be to the intervention groups on the uninvolved side. Patients will present to physical therapy 2-3 times/week during the duration of the study regardless of their group allocation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Diagnosed with rotator cuff injury
* Scheduled for rotator cuff surgery via shoulder arthroscopy

Exclusion Criteria:

* Less than 18 years old
* History of previous contra-lateral surgery or injury
* Previous ipsi-lateral upper extremity surgery
* History of shoulder osteoarthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Change in strength of the shoulder at 6 weeks and 12 weeks | pre-operative visit, 6 week post-operative visit, 12-week post-operative visit
  Strength of the shoulder will be assessed via hand-held dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Banffy, MD, Principal Investigator — Cedars-Sinai Kerlan-Jobe Institute
Locations (1):
- Cedars-Sinai Kerlan-Jobe Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for 6 months after the study has been published.